CLINICAL TRIAL: NCT01500941
Title: Evaluation of the Effects of a Combination of Probiotics in the Treatment of Adult Atopic Dermatitis: Randomized Phase III, Double-blind Placebo-controlled
Brief Title: Probiotics in Adults: do They Improve Atopic Dermatitis?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Iemoli Enrico, head allergy and clinical immunology departement, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 131/2010/77/2009/AP
Record Dates: First submitted 2011-12-21; First posted 2011-12-29 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Adult Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotics (Active Comparator)
  Interventions: Dietary Supplement: probiotics
- maltodextrin (Placebo Comparator)
  Interventions: Other: maltodextrin

INTERVENTIONS:
Dietary Supplement: probiotics — a mixture of Lactobacillus LS01 DSM 2275 and Bifidobacterium BR03 DSM 16604 at a dose of 1 x 109 colony forming units (CFU)/g each in maltodextrin
  Arms: probiotics
Other: maltodextrin — sachets
  Arms: maltodextrin

SUMMARY:
Probiotics are suggested to have beneficial effects in atopic dermatitis (AD) treatment and prevention but their precise role is not yet clear.

The aim of this randomized double blinded active treatment vs placebo study was to evaluate clinical efficacy of intake of a combination of two probiotics (Lactobacillus salivarius LS01 and Bifidobacterium breve BR03) for the treatment of adult AD patients.

The rationale for the use of probiotics in the treatment of atopic dermatitis would be due to some experimental hypotheses:

1. The use of these microbial agents at an early age seems to play an important role in inducing immunity T type 1 (Th1) and inhibit the development of a Th2 response IgE mediated
2. the normal intestinal flora (including probiotics) would play an important role in inducing immunological tolerance
3. the hygiene hypothesis that the reduced bacterial environment would favour a type 2 response T and the development of allergic diseases

ELIGIBILITY:
Inclusion Criteria:Adults aged 18-55 years between

* Diagnosis of DA moderate and / or severe, as assessed by the use of a standardized index of severity of AD (SCORAD = Scoring Atopic Dermatitis index) (42), prepared by the European Task Force for atopic dermatitis

Exclusion Criteria:Allergic contact dermatitis (ACD), active

* In the absence of known food allergy elimination diet
* Chronic diseases (autoimmune diseases, COPD, heart disease, IRC, CNS disease, chronic gastrointestinal diseases, diabetes, congenital or acquired immunosuppression)
* Pregnancy and / or lactation
* Treatment with probiotics in the 6 months preceding enrollment
* Treatment with steroids and antihistamines systemically in the three months prior to enrollment
* Topical treatments with immunomodulators (tacrolimus or pimecrolimus) in the three months prior to enrollment
* Acute or chronic infectious diseases
* Pre-existing hypersensitivity to components contained in the probiotic

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
clinical effects of probiotics on adult atopic dermatitis | 20 weeks
  To evaluate the clinical course of adult patients affected by atopic dermatitis after the intake of two probiotics vs placebo

SECONDARY OUTCOMES:
effects of probiotics on immune system and faecal microbiota in adult atopic dermatitis | 20 weeks
  to evaluate these parameters: percentage of circulating Treg cells, percentage of Th17 cells, Th1 and Th2, percentage of Treg cells TLR2+, TLR4 + and TLR9 +, Quantization plasma LPS. Determination by gene amplification and culture of Lactobacillus salivarius and Bifidobacterium in the faeces of the two groups studied

CONTACTS AND LOCATIONS:
Overall Officials: lorenzo drago, prof, Study Director — Microbiology, Department of Clinical Sciences L. Sacco, University of Milan; 5Laboratory of Clinical Chemistry and Microbiology, IRCCS Galeazzi Orthopaedic Institute, Milan, Italy
Locations (1):
- Luigi Sacco Hospital, Milan, Italy